CLINICAL TRIAL: NCT04399291
Title: A Cross-sectional Analysis of Vitamin D Status and Bone Health of Older Adults Within Residential Care Facilities in Northern Ireland.
Brief Title: Vitamin D Status and Bone Health of Older Adults in Care Facilities
Status: Suspended | Type: Observational
Why Stopped: COVID-19, study status being reviewed on an ongoing basis.
Sponsor: University of Ulster (Other)
Collaborators: Western Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/NI/0114
Record Dates: First submitted 2020-05-11; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Vitamin D Status; Osteoporosis; Sarcopenia
Keywords: Vitamin D; Deficiency; Bone Health; Generic Health Relevance; Musculoskeletal Health; Observation
MeSH Terms: conditions — Osteoporosis; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — White blood, serum, plasma, washed red cells, red cells, buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residential care facility residents: Older adults recruited from care homes in Northern Ireland

SUMMARY:
Vitamin D deficiency is proposed to be prevalent in community-dwelling older adults, with prevalence substantially higher among older adults in residential care facilities. Musculoskeletal health is compromised in older vitamin D deficient individuals and alongside frailty, sarcopenia and osteoporosis associated with ageing, affected individuals are at increased risk of falls and fractures. Vitamin D supplementation is an effective intervention for fall prevention and, along with calcium supplementation, in fracture risk reduction in institutionalised older adults. Thus, monitoring vitamin D status and treating deficiency among older adults in residential care facilities may limit the substantial economic burden associated with falls/fractures in this population. The vitamin D status of older adults in residential care facilities in Northern Ireland (NI) is currently unknown, therefore, the aim of this pilot study is to determine the vitamin D status of this cohort of the population, and to define factors which may influence vitamin D status, including body mass index (BMI), mobility out-of-doors, medication use, dementia and diet. Vitamin D status will be determined via the measurement of 25-hydroxyvitamin D using liquid chromatography-tandem mass spectrometry (LC-MS/MS). In addition, biomarkers associated with vitamin D metabolism will be measured including calcium, albumin, creatinine, urea, bone turnover markers and parathyroid hormone. Factors that may affect vitamin D status will be assessed using a health and lifestyle questionnaire and dietary vitamin D intake will be estimated via analysis of the menus in the residential care facilities. Vitamin D supplementation practices in these facilities will also be assessed via analysis of drug prescription records, focusing on differences between residents who have/have not suffered a fracture. Physical measures such grip strength, timed up and go test and T-score measurement via Achilles ultrasound machine will be taken. This study will provide data on the prevalence of vitamin D deficiency in older adults in residential care facilities within NI and identify factors that predispose residents to increased risk of deficiency. Dissemination of these findings, along with analysis of current supplementation practices, will help practitioners to develop a strategy to identify those residents with vitamin D deficiency/insufficiency and thus requiring supplementation ultimately improving health and well-being. This study will also inform the design of a larger study to investigate vitamin D status, supplementation and musculoskeletal health in older adults in residential care facilities within Northern Ireland, providing important information that will ultimately contribute towards reducing falls and fractures within this population.

ELIGIBILITY:
Inclusion Criteria:

* Currently residing (≥1 month) within a residential care facility in the Western Health and Social Care Trust in Northern Ireland

Exclusion Criteria:

* Participants will be excluded from the study if by the judgement of the consultant rheumatologist that they have very abnormal bone or vitamin D metabolism due to conditions such as end stage renal failure or bone metastases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults within residential care facilities in the Western Health and Social Care Trust in Northern Ireland have been selected to be studied. Residents are being investigated to determine vitamin D status and bone.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Vitamin D status | One day measurement
  25(OH)D status measured by Liquid Chromatography / Mass Spec (LC/MS)

SECONDARY OUTCOMES:
Bone turnover markers | One day measurement
  Osteocalcin, bone-specific alkaline phosphatase
Grip strength | One day measurement
  Measurement taken using hand grip dynamometer
Bone density | One day measurement
  Measured via Achilles heel ultrasound scanner, reported as T-score
Bone Health and lifestyle questionnaire | One day measurement
  General background information related to bone health
Functionality | One day measurement
  Timed up and go test

CONTACTS AND LOCATIONS:
Locations (1):
- Western Health and Social Care Trust care Home facilities, Londonderry, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No